CLINICAL TRIAL: NCT02085382
Title: A Randomized, Controlled Trial of Kangaroo Mother Care in Increasing the Rate of Weight Gain Among Low Birth Weight Neonates Admitted in Level II Neonatal Intensive Care Unit of the Philippine General Hospital
Brief Title: Randomized, Controlled Trial of Kangaroo Mother Care in Increasing the Rate of Weight Gain Among Neonates
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of the Philippines (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NIH 2011-014
Record Dates: First submitted 2014-03-06; First posted 2014-03-12 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-03

CONDITIONS: Low Birth Weight Among Neonates
Keywords: Kangaroo Mother Care(KMC), Low-birth weight, neonates
MeSH Terms: interventions — Kangaroo-Mother Care Method

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Kangaroo Mother Care Group (Other): Mothers in the KMC group were oriented in detail about KMC procedure. The mothers provided skin to skin contact using a specially tailored "kangaroo tube" made of soft flannel cloth. The mothers were encouraged to keep the baby in KMC as long as possible during the day and night for an accumulated time of at least 6 hours per day. The duration of the kangaroo care by each of the mother were recorded and tallied accordingly.
  Interventions: Procedure: Kangaroo Mother Care
- Conventional Mother Care (Other): Conventional method of care was the routine care offered in the neonatal unit to low birth weight infants.
  Interventions: Procedure: Conventional Mother Care

INTERVENTIONS:
Procedure: Kangaroo Mother Care — The infants were placed on continuous skin to skin contact between the mother and the baby as soon as possible. The mother kept her newborn infant between the breast, in close contact with her body and covered with the kangaroo tube. Infants wore diaper and a cap during the procedure. Breastfeeding was the standard feeding method.
  When the baby was not in KMC, the baby was placed in the bassinet under warm lamp, if needed, adequately clothed and covered.
  Arms: Kangaroo Mother Care Group
Procedure: Conventional Mother Care — This is generally included: an artificial warming system (heated room overhead lamp warmers). Breastfeeding was also the standard feeding method but if indicated, babies can also be fed through tube or cup feeding. The mothers were allowed to visit their babies anytime but skin to skin contact was not allowed.
  Babies in both groups were monitored hourly. Their heart rate, respiratory rate and temperature were monitored and recorded. Any untoward events like hypothermia, hypoglycemia, apnea, signs of sepsis, and feeding problems were also noted.
  Arms: Conventional Mother Care

SUMMARY:
A randomized, controlled trial of Kangaroo Mother Care (KMC) to determine the effectiveness in increasing the rate of weight gain among low birth weight neonates.

DETAILED DESCRIPTION:
A randomized, controlled trial of Kangaroo Mother Care (KMC) versus Conventional Care to determine the effectiveness of KMC in increasing the rate of weight gain among low birth weight neonates and if it will decrease sepsis rate and shorten hospital stay among the group.

ELIGIBILITY:
Inclusion Criteria:

* birth weight <1500 grams and stable neonates (no dependency on oxygen and /or intravenous fluid, ability (at least partial) to feed) with stable vital signs for the past 24 hours (normal temperature (36.5-37.5 °C),
* normal heart rate (120-160 bpm), normal blood pressure per age
* no apnea
* no intravenous lines or with well-secured peripheral line
* no sepsis
* no emerging signs of sepsis
* on IV antibiotic therapy but clinically stable
* can require photo therapy but with stable and not rising total serum bilirubin (TSB) level or TSB is not in high risk zone.

Exclusion Criteria:

* neonates with chromosomal and life threatening congenital anomalies, who were severally ill
* whose mothers are critically ill and whose mothers were unable to comply with the follow up schedule.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2011-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Low Birth Weight | 3 days
  Low-birth weight infants both in the intervention and control group were discharged from the study according to the following criteria: baby's general health was good as assessed by the attending physician and in evidence of infection, feeding well and receiving exclusively breast milk, gaining weight (at least 15-20 grams/kg/day for at least 3 days), maintaining body temperature satisfactorily for at least 3 consecutive days in room temperature and the mother and family members were confident to take care of the baby in KMC.

CONTACTS AND LOCATIONS:
Overall Officials: Faye S De Ocampo, Medical Doctor, Principal Investigator — Department of Pediatrics College of Medicine
Locations (1):
- Philippine General Hospital - University of the Philippines Manila, Manila, National Capital Region, Philippines